CLINICAL TRIAL: NCT07171359
Title: Transcranial Magnetic Stimulation (TMS) to Improve Recovery Outcomes Among Patients With Opioid Use Disorder (OUD) and Alcohol Use Disorder (AUD)
Brief Title: TMS to Improve Recovery Outcomes Among Patients With Opioid Use Disorder (OUD) and Alcohol Use Disorder (AUD)
Acronym: TMS4OUDAUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMS4OUDAUD; RECOVERYWORKSNWTMS (Other: RECOVERYWORKSNW)
Record Dates: First submitted 2025-08-26; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Use Disorder; Opioid Use Disorder
Keywords: Transcranial Magnetic Stimulation; Opioid Use Disorder; Alcohol Use Disorder; Intensive Outpatient Treatment; Theta Burst Stimulation
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Treatment As Usual (TAU) for OUD and AUD vs. TAU+TMS 3 minute Theta Burst Stimulation (TBS) vs. TAU+TMS 9 minute TBS, 20 sessions for each individual in the intervention arms over 4 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Treatment As Usual (No Intervention): Study participants in this arm will engage in intensive outpatient alcohol and addiction treatment provided as it usually is for all patients in this program.
- 3-Minute TMS (Active Comparator): TAU + 3-minute TMS: Participants complete TAU as described above, with one 3-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).
  Interventions: Device: TMS Low-Dose
- 9-Minute TMS (Active Comparator): TAU + 9-minute TMS: Participants complete TAU as described above, with one 9-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).
  Interventions: Device: TMS High-Dose

INTERVENTIONS:
Device: TMS Low-Dose — one 3-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).
  Arms: 3-Minute TMS
Device: TMS High-Dose — One 9-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).
  Arms: 9-Minute TMS

SUMMARY:
The study aims to explore the potential of Transcranial Magnetic Stimulation (TMS), particularly Theta Burst Stimulation (TBS), as an adjunctive treatment to enhance recovery outcomes (consumption and craving; withdrawal symptoms; mental, physical, sleep, and cognitive health; engagement with therapy, etc.) in individuals with Opioid Use Disorder (OUD) and individuals with Alcohol Use Disorder (AUD). This project will be completed in partnership with Another Chance Rehab (Portland): Portland's top addiction treatment program offering evidence-based treatment programs for a range of substance use disorders. Another Chance Rehab will serve as the project site for this work.

DETAILED DESCRIPTION:
The investigators will conduct a prospective, randomized, controlled trial. To identify which TMS protocol is most efficacious, there will be three arms to this study.

1. Treatment as Usual (TAU): Participants complete their regularly scheduled therapy activities and receive no add-on TMS. They will answer the demographic survey and outcome measure surveys (listed in a later section).
2. TAU + 3-minute TMS: Participants complete TAU as described above, with one 3-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).
3. TAU + 9-minute TMS: Participants complete TAU as described above, with one 9-minute session of TMS TBS delivered each morning, prior to commencement of their regularly scheduled daily therapy activities, for 5 days/week, for a total of four-weeks (20 sessions total).

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Enrolled in the Intensive Outpatient Program at Another Chance Drug & Alcohol Rehab Center of Portland, Portland, OR.
* Diagnosed with Opioid Use Disorder
* Diagnosed with Alcohol Use Disorder

Exclusion Criteria:

* Children <18 years old
* Pregnant
* Non-English speaking
* Currently taking prescription benzodiazepines or anti-convulsive medications
* In active alcohol or opioid withdrawal
* History of seizure disorder diagnosis
* History of Schizophrenia, Bipolar Disorder, Mania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Engagement in Treatment As Usual activities | 4 weeks
  The Investigators will compare engagement in treatment as usual within and between groups by Number of Days in attendance from baseline assessment to follow up.
Engagement in Treatment As Usual Activities | 4 weeks
  Number of individual treatment sessions attended from baseline assessment to follow up.
Engagement in Treatment As Usual Activities | 4 weeks
  Number of group treatment sessions attended from baseline assessment to follow up.
Engagement in Treatment As Usual Activities | 4 weeks
  Number of negative urine toxicology screens for illicit drugs or unprescribed medications from baseline assessment to follow up.

SECONDARY OUTCOMES:
Delay Discounting | 4 weeks
  On this computer task, participants complete 5 trials where they are asked to choose between an immediate or a delayed reward (e.g., $5 now or $10 in 3 weeks). In this version of the delay discounting task, the delay duration adjusts depending on participants' choice on the previous trial. If participants choose the immediate reward, the next trial will have a shorter duration for the delayed reward (e.g., $10 in 1 day); if participants choose the delayed reward, the next trial will have a longer duration for the delayed reward (e.g., $10 in 2 years). Performance on the delay discounting task is measured by calculating the discounting rate, or the rate at which the value of a reward decreases as a function of delay. Higher discounting rates indicate a preference for smaller immediate rewards over larger delayed rewards and is associated with higher impulsivity. (Koffarnus & Bickel, 2014)
Go/No-Go Task | 4 weeks
  On this computer task, participants are asked to respond to stimuli by either executing ("go" stimuli) or withholding a response ("no-go" stimuli). More "go" stimuli are presented than "no-go" stimuli to induce a prepotent response. Performance on the Go/No-Go task is measured by calculating the proportion of commission errors (i.e., false alarms, making a response to a "no-go" stimulus), omission errors (i.e., misses, failing to respond to a "go" stimulus), and the response times to "go" stimuli. Higher proportions of commission errors are indicative of an inability to inhibit a response, sometimes referred to as rapid-response impulsivity. (Donders, 1969)
Balloon Analogue Risk Task | 4 weeks
  On this computer task, participants are shown a balloon and told that each press of a button will increase the size of the balloon and reward them with a small, hypothetical monetary reward. However, after a variable number of pumps, the balloon will explode, causing them to lose all accumulated rewards on that trial. Participants can pump up the balloon as much as they want before moving onto the next trial. Performance on the BART is measured by calculating the average number of pumps on each balloon excluding balloons that exploded. A higher average number of pumps is associated with more impulsiveness. (BART; Lejuez et al., 2002)
Barratt Impulsiveness Scale-11 | 4 weeks
  On this 30-item questionnaire, participants use a 4-point Likert-type scale (1 = Rarely/Never, 4 = Almost Always/Always) to indicate how frequently statements like "I do things without thinking" and "I concentrate easily" apply to themselves. The BIS-11 total score is a summed score of all responses and can range from 30 to 120, with higher scores indicating higher levels of impulsiveness. There is also an option to calculate scores for three aspects of impulsiveness: attentional, motor, and nonplanning. These subscale scores are calculated by summing the number of associated items. The attentional impulsiveness subscale consists of 8 items, and total scores can range from 8 to 32; the other two subscale scores are 11 items each and scores can range from 11 to 44. (BIS-11; Patton et al., 1995)
Sensation Seeking Scale | 4 weeks
  On this 40-item questionnaire, participants are shown two choices, like "A. I prefer friends who are excitingly unpredictable or B. I prefer friends who are reliable and predictable," and asked to select the statement that most or best describes how they feel. One point is given for the more sensation-seeking choice. The SSS total score is the sum of all more sensation-seeking choices and can range from 0 to 40, with higher scores indicating more sensation-seeking. There is also an option to calculate scores for each of the four factors that make up sensation-seeking: [social and sexual] disinhibition, boredom susceptibility, thrill and adventure seeking, and experience seeking. Each of these scales is made up of 10 of the items and scores can range from 0 to 10. (SSS; Zuckerman et al., 1964)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew E Layton, MD, PhD, Principal Investigator — Washington State University
Locations (1):
- Another Chance Drug & Alcohol Rehab Center of Portland, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
The investigators plan to implement a Data Use and Sharing Agreement between WSU and Another Chance Rehab Center for internal use and collaboration among study team members only. Data collected for this study will be de-identified prior to analysis and dissemination of results, therefore no IPD will be shared with other researchers.

REFERENCES:
- [Background] Liu X, Zhao X, Liu T, Liu Q, Tang L, Zhang H, Luo W, Daskalakis ZJ, Yuan TF. The effects of repetitive transcranial magnetic stimulation on cue-induced craving in male patients with heroin use disorder. EBioMedicine. 2020 Jun;56:102809. doi: 10.1016/j.ebiom.2020.102809. Epub 2020 Jun 5. PMID 32512513
- [Background] Bormann NL, Oesterle TS, Arndt S, Karpyak VM, Croarkin PE. Systematic review and meta-analysis: Combining transcranial magnetic stimulation or direct current stimulation with pharmacotherapy for treatment of substance use disorders. Am J Addict. 2024 May;33(3):269-282. doi: 10.1111/ajad.13517. Epub 2024 Jan 25. PMID 38273429
- [Background] Tsai TY, Wang TY, Liu YC, Lee PW, Chang WH, Lu TH, Tseng HH, Lee SY, Chang YH, Yang Y, Chen PS, Chen KC, Yang YK, Lu RB. Add-on repetitive transcranial magnetic stimulation in patients with opioid use disorder undergoing methadone maintenance therapy. Am J Drug Alcohol Abuse. 2021 May 4;47(3):330-343. doi: 10.1080/00952990.2020.1849247. Epub 2021 Jan 10. PMID 33426970